CLINICAL TRIAL: NCT07161180
Title: A Phase 1 Clinical Trial to Evaluate the Pharmacokinetic Characteristics of "PBK_M2301" in Healthy Adult Volunteers
Brief Title: Evaluation of the Pharmacokinetics of "PBK_M2301" in Healthy Adults
Acronym: PBK_M2301_BE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmbio Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: PBK_M2301_102; PBK_M2301_102 (Other: Pharmbio Korea)
Record Dates: First submitted 2025-08-20; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinetics
MeSH Terms: interventions — dipropizine

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized, two-period, two-sequence crossover study in 32 healthy adult volunteers. Participants will receive a single oral dose of PBK_M2301 or a combination of two reference drugs (R1_PBK_M2301 and R2_PBK_M2301) in a randomized order, with a one-week washout between treatments.
Masking Description: This is an open-label study. No parties, including participants, investigators, care providers, or outcome assessors, are masked to treatment assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: R1_PBK_M2301 + R2_PBK_M2301 Followed by PBK_M2301 (Active Comparator): Participants in this arm will receive a single oral dose of R1_PBK_M2301 (levodropropizine 60 mg) plus R2_PBK_M2301 (Pelargonium sidoides extract 20 mg) in Period 1, followed by a one-week washout, and then a single oral dose of PBK_M2301 (levodropropizine 60 mg + Pelargonium sidoides extract 20 mg) in Period 2. All doses will be administered after at least 10 hours of fasting, with 150 mL of water at room temperature.
  Interventions: Drug: PBK_M2301 (levodropropizine + Pelargonium sidoides extract); Drug: R1_PBK_M2301 (levodropropizine); Drug: R2_PBK_M2301 (Pelargonium sidoides extract)
- Arm 2: PBK_M2301 Followed by R1_PBK_M2301 + R2_PBK_M2301 (Experimental): Participants in this arm will receive a single oral dose of PBK_M2301 (levodropropizine 60 mg + Pelargonium sidoides extract 20 mg) in Period 1, followed by a one-week washout, and then a single oral dose of R1_PBK_M2301 (levodropropizine 60 mg) plus R2_PBK_M2301 (Pelargonium sidoides extract 20 mg) in Period 2. All doses will be administered after at least 10 hours of fasting, with 150 mL of water at room temperature.
  Interventions: Drug: PBK_M2301 (levodropropizine + Pelargonium sidoides extract); Drug: R1_PBK_M2301 (levodropropizine); Drug: R2_PBK_M2301 (Pelargonium sidoides extract)

INTERVENTIONS:
Drug: PBK_M2301 (levodropropizine + Pelargonium sidoides extract) — A single oral tablet containing levodropropizine 60 mg and Pelargonium sidoides extract (11% ethanol dried extract, 5.5~6.6→1) 20 mg. Administered after at least 10 hours of fasting with 150 mL of water at room temperature.
  Other Names: PBK_M2301
Drug: R1_PBK_M2301 (levodropropizine) — A single oral tablet containing levodropropizine 60 mg. Administered after at least 10 hours of fasting with 150 mL of water at room temperature.
  Other Names: R1_PBK_M2301
Drug: R2_PBK_M2301 (Pelargonium sidoides extract) — A single oral tablet containing Pelargonium sidoides extract (11% ethanol dried extract, 5.5~6.6→1) 20 mg. Administered after at least 10 hours of fasting with 150 mL of water at room temperature.
  Other Names: R2_PBK_M2301

SUMMARY:
The goal of this Phase 1 clinical trial is to evaluate the safety and pharmacokinetic characteristics of PBK_M2301 in healthy adult volunteers. The main questions it aims to answer are:

What are the maximum concentration (Cmax) and total drug exposure (AUCt) of PBK_M2301 compared to the combination of two reference drugs?

Are there any safety concerns associated with a single oral dose of PBK_M2301?

Researchers will compare PBK_M2301 with the combination of R1_PBK_M2301 and R2_PBK_M2301 to assess differences in drug levels.

Participants will:

Receive each treatment once in a randomized sequence with a one-week washout in between

Provide blood samples at multiple time points after dosing

Undergo safety assessments including adverse event monitoring, vital signs, laboratory tests, and ECGs

DETAILED DESCRIPTION:
This Phase 1, open-label, randomized, two-period, two-sequence crossover study will evaluate the safety and pharmacokinetic characteristics of PBK_M2301 in 32 healthy adults. PBK_M2301 contains levodropropizine 60 mg and Pelargonium sidoides extract 20 mg per tablet.

Participants will receive either a single dose of PBK_M2301 or a combination of two reference drugs (R1_PBK_M2301 and R2_PBK_M2301) in a randomized sequence, with a one-week washout between treatments. Blood samples will be collected at multiple time points up to 12 hours post-dose to determine plasma concentrations of levodropropizine using a validated LC-MS/MS method.

Primary endpoints are Cmax and AUCt, with secondary endpoints including AUC∞, Tmax, t1/2, CL/F, and Vz/F. Safety will be assessed by monitoring adverse events, vital signs, laboratory tests, and ECGs throughout the study.

ELIGIBILITY:
1 Inclusion Criteria

Subjects who meet all of the following criteria may be included in the study:

1. Male or female subjects aged 19 years or older and less than 65 years at the time of screening.
2. Body mass index (BMI) between 18 and 30 kg/m² (inclusive) at screening (BMI = weight (kg) / height (m)²):

   * For male subjects: body weight ≥ 50 kg.
   * For female subjects: body weight ≥ 45 kg.
3. No clinically significant congenital or chronic diseases, and no pathological symptoms or findings based on internal medicine examination (including, if necessary, electroencephalography, electrocardiography, chest and/or upper gastrointestinal endoscopy, or gastrointestinal radiographic examination).
4. Judged by the principal investigator (or a sub-investigator) to be suitable for participation based on diagnostic tests performed according to the characteristics of the investigational product, including hematology, clinical chemistry, coagulation, serology, urinalysis, and electrocardiography (ECG).
5. Voluntarily decides to participate after receiving and fully understanding a detailed explanation of the study, and signs the written informed consent form, agreeing to comply with the study requirements during the study period.
6. Agrees to use medically acceptable contraception* (excluding hormonal contraceptives) from the first administration of the investigational product until 1 week after the last administration, to prevent pregnancy in themselves or their spouse/partner, and agrees not to donate sperm or ova during this period.

   * Medically acceptable contraception: intrauterine device (IUD), intrauterine system (IUS), vasectomy, tubal ligation, or a combination of barrier methods (male condom, female condom, cervical cap, diaphragm, contraceptive sponge). When using spermicide, at least two barrier methods should be used in combination.

     2 Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from the study:

1. Use of enzyme-inducing or enzyme-inhibiting drugs such as barbiturates within 30 days prior to the first administration, or use of any drugs that may interfere with the study within 10 days prior to the first administration.
2. Participation in a bioequivalence study or any other clinical trial and administration of an investigational product within 6 months prior to the first administration in this study.
3. Whole blood donation within 8 weeks, component blood donation within 2 weeks, or receipt of a blood transfusion within 4 weeks prior to the first administration in this study.
4. History of gastrointestinal resection surgery that may affect drug absorption (excluding appendectomy or hernia repair).
5. Within 1 month prior to the first administration:

   * For male subjects: average alcohol consumption > 21 units/week.
   * For female subjects: average alcohol consumption > 14 units/week.

     (1 unit = 50 mL soju, 250 mL beer, or 30 mL whisky)
   * Average smoking > 20 cigarettes/day.
6. Presence of the following conditions:

   * Known hypersensitivity to the investigational product or any of its components.
   * Bronchial hypersecretion.
   * Mucociliary dysfunction (e.g., Kartagener syndrome, primary ciliary dyskinesia).
   * Increased bleeding tendency or use of anticoagulant therapy.
   * Severe hepatic impairment.
   * Severe liver disease or severe renal disease.
   * Hereditary problems such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
7. History of clinically significant psychiatric disorders.
8. Any other reason, not specified in the inclusion/exclusion criteria, that in the opinion of the principal investigator (or a sub-investigator) makes the subject unsuitable for participation.
9. For female subjects: pregnant, suspected of being pregnant, or breastfeeding.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of Levodropropizine | Pre-dose (0 hours) to 12 hours post-dose (depending on dosing regimen)
  Cmax will be determined from plasma concentration-time data following single and multiple oral doses of PBK_M2301, administered alone and in combination with R1_PBK_M2301 or R2_PBK_M2301.
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration (AUCt) of Levodropropizine | Pre-dose (0 hours) to 12 hours post-dose (depending on dosing regimen)
  AUCt will be calculated using the linear trapezoidal method based on plasma concentration-time data, in accordance with "Regulations on Bioequivalence Tests" (Article 17).

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve extrapolated to infinity (AUC∞) of Levodropropizine | Pre-dose (0 hours) to last quantifiable concentration plus extrapolated terminal phase (up to 12 hours post-dose)
  AUC∞ will be derived as the sum of AUCt and the extrapolated terminal area (Ct/λZ) using noncompartmental analysis, following single and multiple oral doses of Levodropropizine, administered alone and in combination with R1_PBK_M2301 or R2_PBK_M2301.
Ratio of AUCt to AUC∞ of Levodropropizine | Pre-dose (0 hours) to last quantifiable concentration plus extrapolated terminal phase (up to 12 hours post-dose)
  The percentage of AUCt relative to AUC∞ will be calculated for each participant to assess the proportion of the observed exposure, following single and multiple oral doses of Levodropropizine, administered alone and in combination with R1_PBK_M2301 or R2_PBK_M2301.
Time to reach maximum plasma concentration (Tmax) of Levodropropizine | Pre-dose (0 hours) to 12 hours post-dose
  Tmax will be recorded as the actual observed time of maximum plasma concentration for each participant after single and multiple oral doses of Levodropropizine, administered alone and in combination with R1_PBK_M2301 or R2_PBK_M2301.
Terminal elimination half-life (t1/2) of Levodropropizine | From Cmax to terminal phase (up to 12 hours post-dose)
  t1/2 will be estimated from the terminal slope of the log-linear portion of the plasma concentration-time curve after single and multiple oral doses of Levodropropizine, administered alone and in combination with R1_PBK_M2301 or R2_PBK_M2301.
Apparent oral clearance (CL/F) of Levodropropizine | From dosing to terminal phase (up to 12 hours post-dose)
  CL/F will be calculated as the ratio of dose to AUC∞ using noncompartmental methods, following single and multiple oral doses of Levodropropizine, administered alone and in combination with R1_PBK_M2301 or R2_PBK_M2301.
Apparent volume of distribution (Vz/F) of Levodropropizine | From dosing to terminal phase (up to 12 hours post-dose)
  Vz/F will be estimated using noncompartmental analysis based on plasma concentration-time data following single and multiple oral doses of Levodropropizine, administered alone and in combination with R1_PBK_M2301 or R2_PBK_M2301.

CONTACTS AND LOCATIONS:
Locations (1):
- H+ Yangji Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to internal policy and data protection regulations. The dataset is limited to a small population of healthy volunteers and is intended solely for internal analysis and regulatory submission.